CLINICAL TRIAL: NCT00386100
Title: A Randomized, Parallel Group, Double-blind, Multi-center Study Comparing the Efficacy and Safety of AVANDAMET and Metformin After 80 Weeks of Treatment.
Brief Title: A Type 2 Diabetes Study of the Longer-Term Glycemic Effect of AVANDAMET vs. Metformin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVT105913
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Results first posted 2011-04-05 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Fasting Plasma Glucose; Dual energy X ray absorptiometry (DXA); Drug-naive; Type 2 diabetes mellitus; Bone Mineral Density; Hyperglycemia; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — rosiglitazone-metformin combination; Disulfiram; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Placebo Comparator): MET began at a total daily dose of 500 mg and could be increased up to a maximum dose of MET 2000 mg. The dose level was to be increased unless a tolerability issue existed at the current dose level.
  Interventions: Drug: Metformin 500 mg (ttd); Drug: Metformin 1000 mg (ttd); Drug: Metformin 1500 mg (ttd); Drug: Metformin 2000 mg (ttd)
- Avandamet (Rosiglitazone maleate/metformin hydrochloride) (Active Comparator): AVM began at a total daily dose of 4 mg/500 mg and could be increased up to a maximum dose of AVM 8 mg/2000 mg
  Interventions: Drug: Avandamet 6 mg/1500 mg (ttd); Drug: Avandamet 4 mg/1000 mg (ttd); Drug: Avandamet 2 mg/500 mg (ttd); Drug: Avandamet 8 mg/ 2000 mg (ttd)

INTERVENTIONS:
Drug: Avandamet 6 mg/1500 mg (ttd) — One 2 mg/ 500 mg capsule will be taken in the AM with the morning meal Two 2 mg/ 500 mg capsules will be taken in the PM with the evening meal
  Arms: Avandamet (Rosiglitazone maleate/metformin hydrochloride)
Drug: Avandamet 4 mg/1000 mg (ttd) — One 2 mg/500 mg capsule will be taken in the AM with the morning meal. One 2 mg/500 mg capsule will be taken in the PM with the evening meal.
  Arms: Avandamet (Rosiglitazone maleate/metformin hydrochloride)
Drug: Avandamet 2 mg/500 mg (ttd) — one placebo capsule will be taken in the AM with the morning meal one 2 mg/ 500 mg capsule will be taken in the PM with the evening meal.
  Arms: Avandamet (Rosiglitazone maleate/metformin hydrochloride)
Drug: Avandamet 8 mg/ 2000 mg (ttd) — Two 2 mg/ 500 mg capsules will be taken in the AM with the morning meal. Two 2 mg/ 500 mg capsules will be taken in the PM with the evening meal.
  Arms: Avandamet (Rosiglitazone maleate/metformin hydrochloride)
Drug: Metformin 500 mg (ttd) — One placebo capsule will be taken in the AM with the morning meal. One 500 mg capsule will be taken in the PM with the evening meal.
  Arms: Metformin
Drug: Metformin 1000 mg (ttd) — One 500 mg capsule will be taken in the AM with the morning meal. One 500 mg capsule will be taken in the PM with the evening meal.
  Arms: Metformin
Drug: Metformin 1500 mg (ttd) — One 500 mg capsule will be taken in the AM with the morning meal. Two 500 mg capsules will be taken in the PM with the evening meal.
  Arms: Metformin
Drug: Metformin 2000 mg (ttd) — Two 500 mg capsule will be taken in the AM with the morning meal. Two 500 mg capsule will be taken in the PM with the evening meal.
  Arms: Metformin

SUMMARY:
This study will evaluate the longer-term glycemic effect of two medicines approved for initial treatment of type 2 diabetes. The study consists of a 2 week screening period (2 study visits), followed by an 80 week double-blind treatment period (11 study visits). Also, a sub-study was included to look at changes in bone mineral density (BMD) at the lumbar spine.

DETAILED DESCRIPTION:
This was a phase IV, randomized, double-blind, global, multi-centre study. The study consisted of a 2 week screening period followed by an 80 week double-blind treatment period. Subjects who met all eligibility requirements were randomized in a 1:1 ratio, stratified by country, gender (male and female) and pre-screening HbA1c (≤9% or>9) either to MET or AVM. When the substudy was added, a new randomization was created for the participating centers. Those subjects in the bone sub-study were stratified by country, gender (male, premenopausal female, and postmenopausal female), pre-screening HbA1c (i.e., ≤9%; >9%), and either to MET or AVM.

At randomization, Visit 3 (Week 0), subjects were initiated at Dose Level 1. Treatment with AVM was initiated at a dose of 4 mg/500 mg and titrated up to a maximum total daily dose of AVM 8 mg/2000 mg. Treatment with MET therapy was initiated at a dose of 500 mg and titrated up to a maximum daily dose of 2000mg.

ELIGIBILITY:
Inclusion Criteria:

* The subject provides written informed consent.
* The subject is male or female and 18 to 75 years of age at the time of pre-screening.
* The subject has an established clinical diagnosis of type 2 diabetes according to recommended guidelines (e.g., American Diabetes Association, International Diabetes Federation, World Health Organization, Canadian Diabetes Association, or American Association of Clinical Endocrinologists).
* The subject is currently treated with diet and exercise, and has not taken more than 2 weeks of an anti-diabetic monotherapy or insulin in the past 6 months.
* The subject has a BMI >25 kg/m2 at pre-screening.
* The subject has a Quest HbA1c 7.5% to 10.5% at pre-screening.
* The subject has a fasting capillary blood glucose 126 mg/dL (7mmol/L), as measured by the site staff at week 0.
* If the subject is a pre-menopausal female of child-bearing potential, she agrees to practice acceptable contraceptive measures (e.g. oral birth control pills, Norplant, Depo-Provera, an intrauterine device (IUD), a diaphragm with spermicide or a condom with spermicide, or abstinence) at least 1 month before screening, during the study, and for 30 days after the last dose of study medication is taken
* The subject is able and willing to perform self-monitoring of blood glucose as specified in this protocol.

Exclusion Criteria:

* The subject has taken an oral anti-diabetic monotherapy or insulin for more than 14 days in the past 6 months.
* The subject has presence of clinically significant renal or hepatic disease (serum creatinine 1.5 mg/dL (132.6 mol/L) for males and 1.4 mg/dL (123.8 mol/L) for females): ALT, AST, total bilirubin, or alkaline phosphatase >2.5 times the upper limit of the normal (ULN) reference range.
* The subject has anemia defined by hemoglobin concentration <11g/dL (110g/L) for males or <10g/dL (100g/L) for females.
* Presence of unstable or severe angina, coronary insufficiency or New York Heart Association (NYHA) class III-IV or any congestive heart failure requiring pharmacologic treatment.
* The subject has systolic blood pressure >160 mmHg or diastolic blood pressure >90 mmHg
* The subject has a chronic disease requiring intermittent or chronic treatment with oral, intravenous, or intra-articular corticosteroids (i.e., only use of topical, inhaled or nasal corticosteroids is permitted).
* The subject has acute or chronic metabolic acidosis or a history of diabetic ketoacidosis.
* The subject has a clinically significant abnormality which in the judgment of the investigator makes the subject unsuitable for inclusion in the study (e.g., physical examination, laboratory tests, or electrocardiogram, etc).
* The subject has used an investigational agent within 30 days or 5 half-lives (whichever was longer) prior to pre-screening.
* The subject is a female who is lactating, pregnant, or planned to become pregnant.
* The subject has a prior history of severe edema or a medically serious fluid related event (e.g., heart failure).
* The subject has a history of macular edema.
* The subject has significant hypersensitivity (e.g., difficulty swallowing, difficulty breathing, and tachycardia or skin reaction) to TZDs, biguanides, or compounds with similar chemical structures.
* The subject has a diagnosis of cancer (other than squamous, basal cell, or cervical cancer in-situ) in the past 3 years and is receiving treatment for cancer.
* The subject has a history or suspicion of drug abuse or alcohol abuse within the last 6 months.
* The subject is known to have severe lactose intolerance.
* The subject is not willing to comply with visits and procedures described in the protocol.
* The subject has a disease that may affect bone turnover including, but not limited to: Paget's disease, hypercalcemia, hypocalcemia, hyperparathyroidism, hyperthyroidism, osteomalacia, metastatic bone disease
* The subject has a weight of greater than 300 lbs (136.4 kg).
* The subject has received treatment with bisphosphonates (≥1 month cumulative treatment within the last 12 months) or fluoride (dose greater than 10mg/day within the previous 5 years).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Actual)
Dates: Start 2006-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (109):
- United States (68):
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Alhambra, California
  - GSK Investigational Site, Artesia, California
  - GSK Investigational Site, Greenbrae, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Kahului, Hawaii
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Avon, Indiana
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Waterloo, Iowa
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Elkridge, Maryland
  - GSK Investigational Site, Chaska, Minnesota
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, City of Saint Peters, Missouri
  - GSK Investigational Site, Excelsior Springs, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Pahrump, Nevada
  - GSK Investigational Site, Hamilton, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, East Syracuse, New York
  - GSK Investigational Site, Flushing, New York
  - GSK Investigational Site, Kingston, New York
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, Canal Fulton, Ohio
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Mogadore, Ohio
  - GSK Investigational Site, Wandsworth, Ohio
  - GSK Investigational Site, Oregon City, Oregon
  - GSK Investigational Site, Beaver, Pennsylvania
  - GSK Investigational Site, Clairton, Pennsylvania
  - GSK Investigational Site, Coatsville, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Sewickley, Pennsylvania
  - GSK Investigational Site, West Chester, Pennsylvania
  - GSK Investigational Site, Clinton, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Pelzer, South Carolina
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Georgetown, Texas
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Manassas, Virginia
  - GSK Investigational Site, Salem, Virginia
  - GSK Investigational Site, Gig Harbor, Washington
  - GSK Investigational Site, Graham, Washington
  - GSK Investigational Site, Olympia, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Vancouver, Washington
  - GSK Investigational Site, Wenatchee, Washington
  - GSK Investigational Site, Wauwatosa, Wisconsin
- Argentina (7):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Buenos Aries, Buenos Aires
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Mendoza, Mendoza Province
  - GSK Investigational Site, Buenos Aires
- Brazil (6):
  - GSK Investigational Site, Fortaleza, Ceará
  - GSK Investigational Site, Goiânia, Goiás
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Campinas, São Paulo
  - GSK Investigational Site, São Paulo, São Paulo
  - GSK Investigational Site, Brasília
- Canada (9):
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Bathurst, New Brunswick
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Smiths Falls, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Mexico (4):
  - GSK Investigational Site, Tijuana, Baja California Norte
  - GSK Investigational Site, Durango, Durango
  - GSK Investigational Site, Pachuca, Hidalgo
  - GSK Investigational Site, Monterrey, Nuevo León
- Pakistan (2):
  - GSK Investigational Site, Karachi
  - GSK Investigational Site, Lahore
- Philippines (4):
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Marikina City
  - GSK Investigational Site, Quezon City
- South Korea (4):
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon, Kyonggi-do
  - GSK Investigational Site, Uijeongbu-si, Kyonggi-do
- Taiwan (5):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan Hsien

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Borges JL, Bilezikian JP, Jones-Leone AR, Acusta AP, Ambery PD, Nino AJ, Grosse M, Fitzpatrick LA, Cobitz AR. A randomized, parallel group, double-blind, multicentre study comparing the efficacy and safety of Avandamet (rosiglitazone/metformin) and metformin on long-term glycaemic control and bone mineral density after 80 weeks of treatment in drug-naive type 2 diabetes mellitus patients. Diabetes Obes Metab. 2011 Nov;13(11):1036-46. doi: 10.1111/j.1463-1326.2011.01461.x. PMID 21682834
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: AVT105913 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AVT105913 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AVT105913 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AVT105913 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AVT105913 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AVT105913 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AVT105913 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Beginning dose of Metformin (MET) 500 milligrams (mg) once a day. Dose could be increased up to a maximum dose of MET 2000 mg.
- Avandamet: Beginning dose of Avandamet (AVM) 4 mg/500 mg once a day. Dose could be increased up to a maximum dose of 8 mg/2000 mg.
Period: Overall Study
Arm/Group | Metformin | Avandamet
Started | 340 | 348
Completed | 186 | 217
Not Completed | 154 | 131
Not completed — Did not receive study medication | 6 | 4
Not completed — Adverse Event | 15 | 25
Not completed — Death | 0 | 1
Not completed — Insufficient therapeutic effect | 30 | 6
Not completed — Lost to Follow-up | 29 | 29
Not completed — Non-compliance | 18 | 19
Not completed — Protocol Violation | 5 | 3
Not completed — Withdrawal by Subject | 32 | 31
Not completed — Bone mass density (BMD) loss >6% | 4 | 4
Not completed — BMD <2.5 | 1 | 0
Not completed — Consecutive elevated Hba1C | 1 | 0
Not completed — Visit 11 DXA showed excessive bone loss | 0 | 1
Not completed — Laboratory findings | 1 | 0
Not completed — Participant's concern due to CPK levels | 1 | 0
Not completed — Participant moving out of state | 2 | 0
Not completed — Excessive bone loss vs. baseline value | 0 | 1
Not completed — Didn't meet entry criteria | 1 | 1
Not completed — Participant's PCP wanted to stop drug | 1 | 0
Not completed — Osteoporosis findings on Visit 2 DXA | 0 | 1
Not completed — Bad metabolic control & patient security | 1 | 0
Not completed — Bone loss by DXA bone scan | 1 | 0
Not completed — DBP 93 mmHg at randomization | 1 | 0
Not completed — 7.6% bone loss | 1 | 0
Not completed — Osteoporosis | 0 | 1
Not completed — Positive pregnancy test | 1 | 3
Not completed — Out of country for 5 months | 1 | 0
Not completed — Hb1Ac >8% | 0 | 1
Not completed — Participant randomized in error | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Avandamet | Total
Number analyzed (Participants) | 334 | 344 | 678
Age, Continuous [Mean (Standard Deviation); unit: years] — The Safety Population, comprised of all participants who were randomized and received at least one dose of the study medication, was used for all baseline characteristics.
  years | 50.7 (10.49) | 51.5 (10.52) | 51.1 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 160 | 318
  Male | 176 | 184 | 360
Race/Ethnicity, Customized [Number; unit: participants]
  African America/African | 13 | 17 | 30
  American Indian or Alaskan Native | 3 | 7 | 10
  Asian - Central/South Asian | 23 | 22 | 45
  Asian - East Asian | 44 | 51 | 95
  Asian - Japanese | 0 | 1 | 1
  Asian - South East Asian | 48 | 48 | 96
  White - Arabic/North African | 4 | 3 | 7
  White - White/Caucasian/European | 185 | 183 | 368
  Mixed Race | 5 | 5 | 10
  Not Specified | 9 | 7 | 16
Duration of Diabetes [Mean (Standard Deviation); unit: years] — The Safety Population, comprised of all participants who were randomized and received at least one dose of the study medication, was used for all baseline characteristics.
  years | 2.570 (3.2671) | 2.293 (3.0774) | 2.429 (3.1729)

OUTCOME MEASURES:

1. Secondary Outcome: Mean Change From Baseline in HbA1c at Week 80
Description: Blood was taken for serum Hb1AC measurements. Change from baseline was calculated as the Week 80 value minus the baseline value, with LOCF from Week 32 for withdrawn participants or missing values.
Time Frame: Baseline and Week 80
Population: Week 32 Evaluable Population with LOCF: a subset of the ITT Population with LOCF starting at Week 32. Only participants with assessment(s) at Week 32 or later were included in this population. Only evaluable participants, defined as participants with a value at baseline and at the specified visit for the parameter of interest, were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 258 | 265
percent change
  Baseline | 8.59 (0.898) | 8.66 (0.954)
  Change from Baseline | -1.42 (0.070) | -1.91 (0.069)
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment for multiple comparisons; ANCOVA with terms for treatment, region, gender, and baseline value with LOCF from Week 32 for withdrawn participants or missing values; Mean Difference (Net) = -0.49, 95% CI 2-sided [-0.669 to -0.305] — AVM mean change from baseline minus MET mean change from baseline based on ANCOVA model

2. Primary Outcome: Change From Baseline in HbA1c at Week 80
Description: Blood was taken for serum HbA1c measurements. Change from baseline was calculated as the Week 80 value minus the baseline value. Last observation carried forward (LOCF) was not used for this analysis.
Time Frame: Baseline and Week 80
Population: Intent-to-Treat (ITT) Population: all participants who were randomized, received at least one dose of study medication, and had both a baseline and at least one on-therapy value. Only evaluable participants, defined as the number of participants with a baseline and at least one post baseline assessment, were analyzed.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 294 | 301
percent change
  Baseline | 8.64 (0.053) | 8.64 (0.055)
  Change from Baseline | -1.36 (0.073) | -1.85 (0.070)
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p < 0.0001, Repeated measures analysis — No adjustment for multiple comparisons; Repeated measures analysis with terms for baseline, region, treatment, gender, time, and treatment by time interaction; Mean Difference (Net) = -0.50, 95% CI 2-sided [-0.69 to -0.30] — AVM mean change from baseline minus MET mean change from baseline based on repeated measures analysis model

3. Secondary Outcome: Number of Participants Achieving HbA1c <=6.5% and <7% at Week 80
Description: Blood was taken for serum Hb1AC measurements. Hb1AC responders were described as participants having achieved Hb1AC <=6% and <7% at Week 80 with LOCF from Week 32.
Time Frame: Week 80
Population: Week 32 Evaluable Population with LOCF. Only evaluable participants, defined as participants with a value at baseline and at the specified visit for the parameter of interest, were analyzed.
Measure: Number; unit: participants
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 258 | 265
participants
  <=6.5% | 97 | 128
  <7% | 133 | 184
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0046, Regression, Logistic — Hb1AC <= 6.5%; Logistic reggression with terms for treatment, region, gender, and baseline Hb1AC with LOCF from Week 32; Odds Ratio (OR) = 1.18, 95% CI 2-sided [1.18 to 2.46] — Odds of having an HbA1c <= 6.5% at Week 80 on Avandamet compared to Metformin
Statistical Analysis 2: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Hb1AC < 7%; Logistic reggression with terms for treatment, region, gender, and baseline Hb1AC with LOCF from Week 32; Odds Ratio (OR) = 2.59, 95% CI 2-sided [1.75 to 3.81] — Odds of having an HbA1c <7% at Week 80 on Avandamet compared to Metformin

4. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline at Week 80
Description: Blood was taken for serum FPG measurements. Change from baseline was calculated as the Week 80 value minus the baseline value.
Time Frame: Baseline and Week 80
Population: ITT Population. Only evaluable participants, defined as the number of participants with a baseline and at least one post baseline assessment, were analyzed. Last observation carried forward (LOCF) was not used for this analysis.
Measure: Mean (Standard Error); unit: millimoles per Liter (mmol/l)
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 319 | 332
millimoles per Liter (mmol/l)
  Baseline | 10.52 (0.184) | 10.17 (0.162)
  Change from Baseline | -2.25 (0.147) | -3.41 (0.139)
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p < 0.0001, Repeated measures analysis; Terms for baseline, region, treatment, pre-screening Hb1Ac strata, gender, time, and treatment by time interaction; Mean Difference (Net) = -1.15, 95% CI [-1.54 to -0.77] — AVM mean change from baseline minus MET mean change from baseline based on repeated measures analysis model

5. Secondary Outcome: Change From Baseline in FPG at Week 80
Description: Blood was taken for serum FPG measurements. Change from baseline was calculated as the Week 80 value minus the baseline value with LOCF from Week 32 for withdrawn participants or missing values.
Time Frame: Baseline and Week 80
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 258 | 265
mmol/l
  Baseline | 10.37 (3.268) | 10.13 (2.927)
  Change from Baseline | -2.53 (3.165) | -3.39 (2.908)
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for multiple comparisons; Terms for treatment, region, gender, pre-screening Hb1Ac strata, and baseline with LOCF from Week 32 for withdrawn participants or missing values; Median Difference (Net) = -1.07, 95% CI 2-sided [-1.425 to -0.710] — AVM mean change from baseline minus MET mean change from baseline based on ANCOVA model

6. Secondary Outcome: Number of Participants Achieving FPG <=6 mmol/L (110 mg/dL) and <=7 mmol/L (126 mg/dL) at Week 80
Description: Blood was taken for serum FPG measurements. FPG responders were described as participants having achieved FPG <=6 mmol/L (110 mg/dL) and <7 mmol/L (126 mg/dL) Hb1AC at Week 80 with LOCF from Week 32.
Time Frame: Week 80
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 258 | 265
participants
  FPG <=6.1 mmol/l | 31 | 83
  FPG <=7.0 mmol/l | 55 | 133
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — FPG <=6.1 mmol/l; Terms for treatment, region, gender, pre-screening Hb1Ac strata, and baseline with LOCF from Week 32; Odds Ratio (OR) = 4.47, 95% CI 2-sided [2.94 to 6.81] — Odds of having an FPG <=6.1 mmol/l at Week 80 on Avandamet compared to Metformin
Statistical Analysis 2: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — FPG <=7 mmol/l; Terms for treatment, region, gender, pre-screening Hb1Ac, and baseline with LOCF from Week 32; Odds Ratio (OR) = 3.33, 95% CI 2-sided [2.25 to 4.92] — Odds of having an FPG <=7 mmol/l at Week 80 on Avandamet compared to Metformin

7. Secondary Outcome: Number of Participants Achieving Treatment Failure
Description: Treatment failure was defined as an HbA1c level >= 7% after Week 32 or withdrawal due to insufficient therapeutic effect (ITE) at any time.
Time Frame: Randomization to treatment failure (up to Week 80)
Population: ITT Population. Only evaluable participants, defined as the number of subjects with a baseline and at least one post baseline assessment, were analyzed. Last observation carried forward (LOCF) was not used for this analysis
Measure: Number; unit: participants
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 319 | 332
participants | 156 | 114
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Cox proportional hazard regression with terms for treatment, region, baseline Hb1Ac strata, and gender; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.45 to 0.74]

8. Secondary Outcome: Percent Change From Baseline in Total Cholesterol, Low-density Lipoprotein (LDL) Cholesterol, High-density Lipoprotein (HDL) Cholesterol, and Triglycerides at Week 80
Description: Blood was taken for measurement of total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides. Percent change from baseline at Week 80 was based on log transformed data. Geometric mean, GM; standard error, SE. n is the number of evaluable participants, which is the number of participants with a value at baseline and at the specified visit for the parameter of interest.
Time Frame: Baseline and Week 80
Population: Week 32 evaluable population with LOCF from Week 32. n is the number of evaluable participants, which is defined as the number of participants with a value at baseline and at the specified visit for the parameter of interest.
Measure: Number; unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 258 | 265
percent change
  % change + SE, Total cholesterol, n=258, 265 | -1.615 | 4.218
  % change, Total cholesterol, n=258, 265 | -2.89 | 2.91
  % change - SE, Total cholesterol, n=258, 265 | -4.140 | 1.614
  % change + SE, LDL cholesterol, n=248, 252 | -4.933 | 3.304
  % change, LDL cholesterol, n=248, 252 | -7.11 | 0.98
  % change - SE, LDL cholesterol, n=248, 252 | -9.228 | -1.286
  % change + SE, HDL cholesterol, n=258, 265 | 6.761 | 9.483
  % change, HDL cholesterol, n=258, 265 | 5.60 | 8.324
  % change - SE, HDL cholesterol, n=258, 265 | 4.453 | 7.179
  % change + SE, triglycerides, n=258, 265 | -2.696 | -2.042
  % change, triglycerides, n=258, 265 | -5.330 | -4.627
  % change - SE, triglycerides, n=258, 265 | -7.893 | -7.143
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0006, ANCOVA — Total cholesterol. No adjustment for multiple comparisons. Log transformed; ANCOVA with log (value) minus log (baseline [BL]) as dependent variable. Terms for treatment, region, gender, pre-screening HbA1c strata, and log (BL); Percent difference from metformin = 5.97, 95% CI 2-sided [2.522 to 9.526]
Statistical Analysis 2: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.056, ANCOVA — LDL cholesterol. No adjustment for multiple comparisons. Log transformed; [statistical method as in outcome 8, analysis 1]; Percent difference from metformin = 8.71, 95% CI 2-sided [2.486 to 15.304]
Statistical Analysis 3: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.072, ANCOVA — HDL cholesterol. No adjustment for multiple comparison. Log transformed; [statistical method as in outcome 8, analysis 1]; Percent difference from metformin = 2.580, 95% CI 2-sided [-0.232 to 5.470]
Statistical Analysis 4: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.835, ANCOVA — Triglycerides. No adjustment for multiple comparisons. Log transformed; [statistical method as in outcome 8, analysis 1]; Percent difference from metformin = 0.743, 95% CI 2-sided [-6.056 to 8.035]

9. Secondary Outcome: Percent Change From Baseline in Adiponectin at Week 80 (United States [US] and Mexico Subset of Participants )
Description: Blood was taken for measurement of adiponectin. Percent change from baseline at Week 80 was based on log transformed data. This outcome measure was analyzed for a subset of participants in the US and Mexico only.
Time Frame: Baseline and Week 80
Population: Week 32 Evaluable Population with LOCF for US and Mexico subset. Only evaluable participants, defined as the number of participants with a value at baseline and at the specified visit for the parameter of interest, were analyzed.
Measure: Number; unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 91 | 96
percent change
  Percent change from baseline + SE | 18.58 | 139.28
  Percent change from baseline | 12.96 | 128.44
  Percent change from baseline - SE | 7.61 | 118.10
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p < 0.0001, ANCOVA — No adjustment for multiple comparisons. Log transformed; [statistical method as in outcome 8, analysis 1]; Percent difference from metformin = 102.24, 95% CI 2-sided [79.23 to 128.19]

10. Secondary Outcome: Percent Change From Baseline in C-reactive Protein (CRP) at Week 80 (US and Mexico Subset of Participants)
Description: Blood was taken for measurement of CRP. Percent change from baseline at Week 80 was based on log transformed data. This outcome measure was analyzed for a subset of participants in the US and Mexico only.
Time Frame: Baseline and Week 80
Population: as for outcome 9
Measure: Number; unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 92 | 95
percent change
  Percent change from baseline + SE | -6.49 | 14.28
  Percent change from baseline | -10.63 | -17.96
  Percent change from baseline - SE | -14.59 | -21.49
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.1380, ANCOVA — No adjustment for multiple comparisons. Log transformed; [statistical method as in outcome 8, analysis 1]; Percent difference from metformin = -8.20, 95% CI 2-sided [-18.04 to 2.82]

11. Secondary Outcome: Percent Change in Free Fatty Acids (FFA) From Baseline at Week 80 (US and Mexico Subset of Participants).
Description: Blood was taken for measurement of FFA. Percent change from baseline at Week 80 was based on log transformed data. This outcome measure was analyzed for a subset of participants in the US and Mexico only.
Time Frame: Baseline and Week 80
Population: Week 32 Evaluable Population with LOCF for US and Mexico subset. Only evaluable participants, defined as participants with a value at baseline and at the specified visit for the parameter of interest, were analyzed.
Measure: Number; unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 92 | 95
percent change
  Percent change from baseline + SE | 14.353 | 1.267
  Percent change from baseline | 9.40 | -2.97
  Percent change from baseline - SE | 4.657 | -7.028
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0342, ANCOVA — No adjustment for multiple comparisons. Log transformed; [statistical method as in outcome 8, analysis 1]; Percent difference from metformin = -11.308, 95% CI 2-sided [-20.617 to -0.899]

12. Secondary Outcome: Change in Fasting Insulin From Baseline at Week 80 (US and Mexico Subset of Participants)
Description: Blood was taken for fasting insulin measurements. Change from baseline was calculated as the Week 80 value minus the baseline value, with LOCF from Week 32 for withdrawn participants or missing values. This outcome measure was analyzed for a subset of participants in the US and Mexico only.
Time Frame: Baseline and Week 80
Population: as for outcome 11
Measure: Mean (Standard Error); unit: picomoles per Liter (pmol/l)
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 92 | 97
picomoles per Liter (pmol/l) | -1.5 (9.18) | -35.2 (8.79)
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0042, ANCOVA — No adjustment for multiple comparisons; ANCOVA with terms for treatment, region, gender, pre-screening HbA1c strata, and baseline; Mean Difference (Net) = -33.7, 95% CI 2-sided [-56.666 to -0.99] — AVM mean change from baseline minus MET mean change from baseline based on ANCOVA model

13. Secondary Outcome: Change in C-peptide From Baseline at Week 80 (US and Mexico Subset of Participants)
Description: Blood was taken for C-peptide measurements. Change from baseline was calculated as the Week 80 value minus the baseline value with LOCF from Week 32 for withdrawn participants or missing values. This outcome measure was analyzed for a subset of participants in the US and Mexico only.
Time Frame: Baseline and Week 80
Population: as for outcome 11
Measure: Mean (Standard Error); unit: mmol/l
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 92 | 95
mmol/l | -0.244 (0.0518) | -0.473 (0.0502)
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0006, ANCOVA — No adjustment for multiple comparisons; ANCOVA with terms for treatment, region, gender, pre-screening HbA1c strata, and baseline; Median Difference (Net) = -0.229, 95% CI 2-sided [-0.359 to -0.099] — AVM mean change from baseline minus MET mean change from baseline based on ANCOVA model

14. Secondary Outcome: Percent Change From Baseline in in HOMA-S and HOMA-B to Week 80 (US and Mexico Subset of Participants)
Description: Blood was taken for measurement of homeostasis model assessment for insulin sensitivity (HOMA-S) and beta-cell function (HOMA-B). Percent change from baseline at Week 80 was based on log transformed data. This outcome measure was analyzed for a subset of participants in the US and Mexico only. GM, geometric mean; SE, standard error.
Time Frame: Baseline and Week 80
Population: as for outcome 11
Measure: Number; unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 91 | 96
percent change
  Percent change HOMA-B + SE | 88.25 | 92.32
  Percent change HOMA-B | 78.85 | 83.14
  Percent change HOMA-B - SE | 69.92 | 74.39
  Percent change HOMA-S + SE | 25.13 | 63.67
  Percent change HOMA-S | 18.65 | 55.58
  Percent change HOMA-S - SE | 12.49 | 47.91
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.7148, ANCOVA — HOMA-B. Log transformed; [statistical method as in outcome 8, analysis 1]; Percent difference from metformin = 2.40, 95% CI 2-sided [-9.87 to 16.34]
Statistical Analysis 2: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p < 0.001, ANCOVA — HOMA-S. Log transformed; [statistical method as in outcome 8, analysis 1]; percent difference from metformin = 31.14, 95% CI 2-sided [14.82 to 49.78]

15. Secondary Outcome: Slope of Delta-cell Function as Estimated by the Ratio deltaI/deltaG
Description: The ratio Delta I/Delta G is calculated based on the oral glucose tolerance test (OGTT), where Delta I = (30 minute immunoreactive insulin minus 0 minute immunoreactive insulin) and Delta G = (30 minute plasma glucose minus 0 minute plasma glucose). The 0 minute values are fasting insulin and glucose; the 30 minute values are taken 30 minutes after the oral glucose challenge. This outcome measure was analyzed for a subset of participants in the US and Mexico only.
Time Frame: Baseline and Week 80
Population: Week 32 Evaluable Population with LOCF. Only evaluable participants, defined as participants from US and Mexico sites with a value at baseline and at the specified visit, were analyzed.
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 82 | 89
ratio | -86.23 (59.706) | -5.38 (55.229)
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.319, Repeated measures analysis; Repeated measures analysis with terms for baseline, region, treatment, gender, pre-screening Hb1AC, time, and treatment by time interaction; Mean Difference (Net) = 80.85, 95% CI 2-sided [-79.035 to 240.744]

16. Secondary Outcome: Number of Participants at Final Dose Level
Time Frame: Baseline to Week 80 or withdrawal
Population: Safety population. This population consisted of all participants who were randomized and received at least one dose of the study medication.
Measure: Number; unit: participants
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 334 | 344
participants
  Dose level 1 AVM 4 mg/500 mg, MET 500 mg | 17 | 19
  Dose level 2 AVM 4 mg/1000 mg, MET 1000 mg | 16 | 18
  Dose level 3 AVM 6 mg/1500 mg, MET 1500 mg | 27 | 34
  Dose level 4 AVM 8 mg/2000 mg, MET 2000 mg | 236 | 242

17. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mass Density (BMD) at Weeks 20, 56, and 80 (Bone Sub-study Subset of Participants)
Description: BMD was measured by dual X-ray absorptiometry (DXA). The percent change from baseline in BMD at a given timepoint was defined at the participant level by the following formula: percent change = (BMD at given week minus BMD at baseline)/BMD at baseline x 100%. This outcome measure was analyzed for a subset of participants in the bone study only.
Time Frame: Baseline and Weeks 20, 56, and 80
Population: Week 20 Evaluable for the Bone Sub-study Population. This is a subset of the bone sub-study with LOCF from Week 20. Only participants with BMD assessment(s) at Week 20 or later were included.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 87 | 87
percent change
  Overall population, Week 80, n=87, 87 | -2.1 (0.54) | 0.1 (0.54)
  Overall population, Week 56, n=87, 87 | -1.4 (0.45) | 0.3 (0.44)
  Overall population, Week 20, n=87, 87 | -0.5 (0.41) | 0.5 (0.40)
  Male population, Week 80, n=38, 43 | -0.7 (0.81) | 1.0 (0.90)
  Male population, Week 56, n=38, 43 | -0.2 (0.61) | 0.7 (0.68)
  Male population, Week 20, n=38, 43 | -0.1 (0.63) | -0.2 (0.71)
  Female population, Week 80, n=49, 44 | -2.7 (0.77) | 0.2 (0.75)
  Female population, Week 56, n=49, 44 | -2.0 (0.70) | 0.3 (0.68)
  Female population, Week 20, n=49, 44 | -0.9 (0.52) | 1.2 (0.51)
  Premenopausal population, Week 80, n=21, 14 | -2.4 (1.01) | -0.7 (1.03)
  Premenopausal population, Week 56, n=21, 14 | -0.8 (0.88) | 0.2 (0.90)
  Premenopausal population, Week 20, n=21, 14 | 0.2 (0.75) | 0.5 (0.77)
  Postmenopausal population, Week 80, n=28, 30 | -3.3 (1.22) | 0 (1.16)
  Postmenopausal population, Week 56, n=28, 30 | -2.7 (1.09) | -0.1 (1.04)
  Postmenopausal population, Week 20, n=28, 30 | -1.4 (0.73) | -1.1 (0.69)
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0012, ANCOVA — Overall population, Week 80. No adjustment for multiple comparisons. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -2.2, 95% CI 2-sided [-3.5 to -0.9]
Statistical Analysis 2: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0031, ANCOVA — Overall population, Week 56. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -1.6, 95% CI 2-sided [-2.7 to -0.6]
Statistical Analysis 3: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0308, ANCOVA — Overall population, Week 20. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -1.1, 95% CI 2-sided [-2.0 to -0.1]
Statistical Analysis 4: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0954, ANCOVA — Male population, Week 80. No adjustment for multiple comparisons. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -1.7, 95% CI 2-sided [-3.7 to 0.3]
Statistical Analysis 5: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0015, ANCOVA — Female population, Week 80. No adjustment for multiple comparisons. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -2.9, 95% CI 2-sided [-4.7 to -1.2]
Statistical Analysis 6: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0045, ANCOVA — Female population, Week 56. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -2.3, 95% CI 2-sided [-3.9 to -0.7]
Statistical Analysis 7: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0005, ANCOVA — Female population, Week 20. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -2.2, 95% CI 2-sided [-3.3 to -1.0]
Statistical Analysis 8: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.2363, ANCOVA — Premenopausal female population, Week 80. No adjustment for multiple comparisons. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -1.7, 95% CI 2-sided [-4.6 to 1.2]
Statistical Analysis 9: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0161, ANCOVA — Postmenopausal female population, Week 80. No adjustment for multiple comparisons. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -3.3, 95% CI 2-sided [-5.9 to -0.6]
Statistical Analysis 10: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0338, ANCOVA — Postmenopausal female population, Week 56. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -2.6, 95% CI 2-sided [-4.9 to -0.2]
Statistical Analysis 11: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0020, ANCOVA — Postmenopausal female population, Week 20. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Median Difference (Net) = -2.6, 95% CI 2-sided [-4.1 to -1.0]

18. Secondary Outcome: Percent Change From Baseline in Total Hip BMD at Weeks 20, 56, and 80 (Bone Sub-study Subset of Participants)
Description: BMD was measured by dual X-ray absorptiometry (DXA). The percent change from baseline in BMD at a given timepoint was defined at the participant level by the following formula: percent change = (BMD at given week minus BMD at baseline)/BMD at baseline x 100. This outcome measure was analyzed for a subset of participants in the bone study only.
Time Frame: Baseline and Weeks 20, 56, and 80
Population: as for outcome 17
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 87 | 87
percent change
  Overall population, Week 80, n=87, 87 | 0.0 (0.35) | -1.5 (0.35)
  Overall population, Week 56, n=87, 87 | -0.2 (0.31) | -1.2 (0.32)
  Overall population, Week 20, n=87, 87 | 0.2 (0.24) | -0.4 (0.24)
  Male population, Week 80, n=38, 43 | 0.3 (0.46) | -1.0 (0.41)
  Male population, Week 56, n=38, 43 | 0.2 (0.41) | -0.8 (0.37)
  Male population, Week 20, n=38, 43 | 0.5 (0.35) | -0.3 (0.31)
  Female population, Week 80, n=49, 44 | 0.0 (0.60) | -1.8 (0.61)
  Female population, Week 56, n=49, 44 | -0.2 (0.52) | -1.4 (0.54)
  Female population, Week 20, n=49, 44 | -0.3 (0.37) | -0.6 (0.38)
  Premenopausal population, Week 80, n=21, 14 | 1.3 (0.71) | -0.9 (0.69)
  Premenopausal population, Week 56, n=21, 14 | 0.8 (0.69) | -1.6 (0.67)
  Premenopausal population, Week 20, n=21, 14 | 0.3 (0.48) | 0.0 (0.47)
  Postmenopausal population, Week 80, n=28, 30 | -0.9 (0.97) | -2.3 (1.02)
  Postmenopausal population, Week 56, n=28, 30 | -1.1 (0.81) | -1.5 (0.85)
  Postmenopausal population, Week 20, n=28, 30 | -0.4 (0.57) | -0.6 (0.60)
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0005, ANCOVA — [p-value comment as in outcome 17, analysis 1]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -1.5, 95% CI 2-sided [-2.3 to -0.7]
Statistical Analysis 2: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0110, ANCOVA — [p-value comment as in outcome 17, analysis 2]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Median Difference (Net) = -1.0, 95% CI 2-sided [-1.7 to -0.2]
Statistical Analysis 3: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0618, ANCOVA — [p-value comment as in outcome 17, analysis 3]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.1 to 0.0]
Statistical Analysis 4: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0110, ANCOVA — [p-value comment as in outcome 17, analysis 4]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -1.3, 95% CI 2-sided [-2.3 to -0.3]
Statistical Analysis 5: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0272, ANCOVA — Male population, Week 56. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -1.0, 95% CI 2-sided [-1.9 to -0.1]
Statistical Analysis 6: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0337, ANCOVA — Male population, Week 20. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -0.8, 95% CI 2-sided [-1.6 to -0.1]
Statistical Analysis 7: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0152, ANCOVA — [p-value comment as in outcome 17, analysis 5]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Median Difference (Net) = -1.7, 95% CI 2-sided [-3.1 to -0.3]
Statistical Analysis 8: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0570, ANCOVA — [p-value comment as in outcome 17, analysis 6]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -1.2, 95% CI 2-sided [-2.4 to 0.0]
Statistical Analysis 9: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0296, ANCOVA — [p-value comment as in outcome 17, analysis 8]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Median Difference (Net) = -2.2, 95% CI 2-sided [-4.3 to -0.2]
Statistical Analysis 10: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0155, ANCOVA — Premenopausal female population, Week 56. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -2.4, 95% CI 2-sided [-4.4 to -0.5]
Statistical Analysis 11: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.5870, ANCOVA — Premenopausal female population, Week 20. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Median Difference (Net) = -0.4, 95% CI 2-sided [-1.7 to 1.0]
Statistical Analysis 12: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.1854, ANCOVA — [p-value comment as in outcome 17, analysis 9]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -1.5, 95% CI 2-sided [-3.6 to 0.7]

19. Secondary Outcome: Percent Change From Baseline in Trochanter BMD at Weeks 20, 56, and 80 (Bone Sub-study Subset of Participants)
Description: as for outcome 18
Time Frame: Baseline and Weeks 20, 56, and 80
Population: as for outcome 17
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 87 | 87
percent change
  Overall population, Week 80, n=87, 87 | -0.1 (0.54) | -2.1 (0.55)
  Overall population, Week 56, n=87, 87 | -0.2 (0.49) | -1.7 (0.49)
  Overall population, Week 20, n=87, 87 | 0.1 (0.35) | -0.6 (0.34)
  Male population, Week 80, n=38, 43 | 1.1 (0.69) | -0.4 (0.61)
  Male population, Week 56, n=38, 43 | 0.9 (0.67) | -0.5 (0.60)
  Male population, Week 20, n=38, 43 | 0.7 (0.55) | -0.2 (0.48)
  Female population, Week 80, n=49, 44 | -0.2 (0.93) | -2.6 (0.96)
  Female population, Week 56, n=49, 44 | -0.3 (0.80) | -2.1 (0.82)
  Female population, Week 20, n=49, 44 | -0.2 (0.52) | -0.8 (0.53)
  Premenopausal population, Week 80, n=21, 14 | 1.7 (1.18) | -1.4 (1.12)
  Premenopausal population, Week 56, n=21, 14 | 0.3 (0.94) | -2.6 (0.89)
  Premenopausal population, Week 20, n=21, 14 | 0.0 (0.71) | 0.0 (0.67)
  Postmenopausal population, Week 80, n=28, 30 | -1.1 (1.45) | -3.6 (1.53)
  Postmenopausal population, Week 56, n=28, 30 | -1.1 (1.25) | -2.2 (1.31)
  Postmenopausal population, Week 20, n=28, 30 | -0.3 (0.76) | -1.0 (0.80)
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0038, ANCOVA — [p-value comment as in outcome 17, analysis 1]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Median Difference (Net) = -1.9, 95% CI 2-sided [-3.2 to -0.6]
Statistical Analysis 2: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0134, ANCOVA — [p-value comment as in outcome 17, analysis 2]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -1.5, 95% CI 2-sided [-2.7 to -0.3]
Statistical Analysis 3: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0967, ANCOVA — [p-value comment as in outcome 17, analysis 3]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Median Difference (Net) = -0.7, 95% CI 2-sided [-1.5 to 0.1]
Statistical Analysis 4: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0512, ANCOVA — [p-value comment as in outcome 17, analysis 4]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -1.5, 95% CI 2-sided [-3.0 to 0.0]
Statistical Analysis 5: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0330, ANCOVA — [p-value comment as in outcome 17, analysis 5]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -2.4, 95% CI 2-sided [-4.6 to -0.2]
Statistical Analysis 6: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0547, ANCOVA — [p-value comment as in outcome 17, analysis 6]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -1.8, 95% CI 2-sided [-3.7 to 0.0]
Statistical Analysis 7: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.0613, ANCOVA — [p-value comment as in outcome 17, analysis 8]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -3.1, 95% CI 2-sided [-6.3 to 0.2]
Statistical Analysis 8: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.1369, ANCOVA — [p-value comment as in outcome 17, analysis 9]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -2.5, 95% CI 2-sided [-3.9 to 1.7]

20. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD at Weeks 20, 56, and 80 (Bone Sub-study Subset of Participants)
Description: as for outcome 18
Time Frame: Baseline and Weeks 20, 56, and 80
Population: as for outcome 17
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 87 | 87
percent change
  Overall population, Week 80, n=87, 87 | -0.7 (0.39) | -1.4 (0.39)
  Overall population, Week 56, n=87, 87 | -0.7 (0.39) | -0.8 (0.39)
  Overall population, Week 20, n=87, 87 | -0.1 (0.36) | -0.2 (0.36)
  Male population, Week 80, n=38, 43 | -1.4 (0.66) | -2.2 (0.59)
  Male population, Week 56, n=38, 43 | -0.7 (0.64) | -1.3 (0.57)
  Male population, Week 20, n=38, 43 | -0.4 (0.60) | -0.7 (0.53)
  Female population, Week 80, n=49, 44 | -0.3 (0.56) | -1.2 (0.57)
  Female population, Week 56, n=49, 44 | -0.6 (0.55) | -0.5 (0.56)
  Female population, Week 20, n=49, 44 | -0.4 (0.49) | -0.2 (0.50)
  Premenopausal population, Week 80, n=21, 14 | 0.9 (0.73) | -0.3 (0.68)
  Premenopausal population, Week 56, n=21, 14 | -0.1 (0.96) | -0.4 (0.89)
  Premenopausal population, Week 20, n=21, 14 | 0.9 (0.83) | -0.3 (0.77)
  Postmenopausal population, Week 80, n=28, 30 | -1.3 (0.87) | -2.1 (0.91)
  Postmenopausal population, Week 56, n=28, 30 | -1.2 (0.81) | -0.7 (0.85)
  Postmenopausal population, Week 20, n=28, 30 | -1.1 (0.71) | -0.4 (0.74)
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.1260, ANCOVA — [p-value comment as in outcome 17, analysis 1]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Median Difference (Net) = -0.7, 95% CI 2-sided [-1.7 to 0.2]
Statistical Analysis 2: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.3117, ANCOVA — [p-value comment as in outcome 17, analysis 4]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Median Difference (Net) = -0.7, 95% CI 2-sided [-2.2 to 0.7]
Statistical Analysis 3: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.1776, ANCOVA — [p-value comment as in outcome 17, analysis 5]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -0.9, 95% CI 2-sided [-2.2 to 0.4]
Statistical Analysis 4: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.2259, ANCOVA — [p-value comment as in outcome 17, analysis 8]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Median Difference (Net) = -1.2, 95% CI 2-sided [-3.2 to 0.8]
Statistical Analysis 5: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.3840, ANCOVA — [p-value comment as in outcome 17, analysis 9]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -0.9, 95% CI 2-sided [-2.8 to 1.1]

21. Secondary Outcome: Percent Change From Baseline in Distal Radius BMD at Weeks 20, 56, and 80 (Bone Sub-study Subset of Participants)
Description: as for outcome 18
Time Frame: Baseline and Weeks 20, 56, and 80
Population: as for outcome 17
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 87 | 87
percent change
  Overall population, Week 80, n=87, 87 | 0.3 (0.63) | -0.1 (0.66)
  Overall population, Week 56, n=87, 87 | 0.5 (0.55) | 0.5 (0.58)
  Overall population, Week 20, n=87, 87 | 1.2 (0.58) | 0.9 (0.61)
  Male population, Week 80, n=38, 43 | 0.4 (0.84) | -0.6 (0.82)
  Male population, Week 56, n=38, 43 | 0.7 (0.73) | 0.4 (0.71)
  Male population, Week 20, n=38, 43 | 1.5 (0.75) | 0.2 (0.73)
  Female population, Week 80, n=49, 44 | 0.1 (1.00) | 0.1 (1.07)
  Female population, Week 56, n=49, 44 | 0.6 (0.87) | 0.7 (0.93)
  Female population, Week 20, n=49, 44 | 0.6 (0.94) | 1.1 (0.99)
  Premenopausal population, Week 80, n=21, 14 | 1.1 (1.51) | -0.3 (1.44)
  Premenopausal population, Week 56, n=21, 14 | 2.2 (1.37) | -0.6 (1.30)
  Premenopausal population, Week 20, n=21, 14 | 2.6 (1.51) | 0.7 (1.40)
  Postmenopausal population, Week 80, n=28, 30 | -0.5 (1.61) | -0.2 (1.76)
  Postmenopausal population, Week 56, n=28, 30 | -0.3 (1.34) | 0.8 (1.46)
  Postmenopausal population, Week 20, n=28, 30 | 0.5 (1.36) | 1.3 (1.49)
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.6102, ANCOVA — [p-value comment as in outcome 17, analysis 1]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.9 to 1.1]
Statistical Analysis 2: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.3445, ANCOVA — [p-value comment as in outcome 17, analysis 4]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -0.9, 95% CI 2-sided [-2.9 to 1.0]
Statistical Analysis 3: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.9735, ANCOVA — [p-value comment as in outcome 17, analysis 5]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = 0.0, 95% CI 2-sided [-2.4 to 2.3]
Statistical Analysis 4: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.4861, ANCOVA — [p-value comment as in outcome 17, analysis 8]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -1.4, 95% CI 2-sided [-5.8 to 2.9]
Statistical Analysis 5: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.8770, ANCOVA — [p-value comment as in outcome 17, analysis 9]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = 0.3, 95% CI 2-sided [-3.5 to 4.0]

22. Secondary Outcome: Percent Change From Baseline in Total Body BMD at Weeks 20, 56, and 80 (Bone Sub-study Subset of Participants)
Description: as for outcome 18
Time Frame: Baseline and Weeks 20, 56, and 80
Population: as for outcome 17
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 87 | 87
percent change
  Overall population, Week 80, n=87, 87 | 1.1 (0.64) | 1.1 (0.64)
  Overall population, Week 56, n=87, 87 | 1.3 (0.63) | -0.1 (0.63)
  Overall population, Week 20, n=87, 87 | 0.0 (0.37) | 0.5 (0.37)
  Male population, Week 80, n=38, 43 | 0.3 (0.43) | 0.5 (0.38)
  Male population, Week 56, n=38, 43 | 0.5 (0.41) | 0.5 (0.37)
  Male population, Week 20, n=38, 43 | 0.2 (0.43) | 0.5 (0.38)
  Female population, Week 80, n=49, 44 | 2.0 (1.00) | 1.0 (1.01)
  Female population, Week 56, n=49, 44 | 1.9 (1.03) | 1.2 (1.04)
  Female population, Week 20, n=49, 44 | -0.2 (0.56) | 0.5 (0.57)
  Premenopausal population, Week 80, n=21, 14 | 5.3 (2.26) | -0.2 (2.73)
  Premenopausal population, Week 56, n=21, 14 | 5.2 (2.42) | -1.0 (2.94)
  Premenopausal population, Week 20, n=21, 14 | -0.2 (1.38) | 0.3 (1.66)
  Postmenopausal population, Week 80, n=28, 30 | 0.2 (0.56) | -0.4 (0.67)
  Postmenopausal population, Week 56, n=28, 30 | -0.2 (0.49) | -0.6 (0.58)
  Postmenopausal population, Week 20, n=28, 30 | -0.2 (0.45) | 0.1 (0.54)
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.7015, ANCOVA — [p-value comment as in outcome 17, analysis 1]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Median Difference (Net) = -0.2, 95% CI 2-sided [-1.5 to 1.0]
Statistical Analysis 2: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.6767, ANCOVA — [p-value comment as in outcome 17, analysis 4]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.7 to 1.0]
Statistical Analysis 3: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.4199, ANCOVA — [p-value comment as in outcome 17, analysis 5]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -1.0, 95% CI 2-sided [-3.4 to 1.5]
Statistical Analysis 4: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.2526, ANCOVA — [p-value comment as in outcome 17, analysis 8]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Median Difference (Net) = -5.5, 95% CI 2-sided [-16.4 to 5.4]
Statistical Analysis 5: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.4153, ANCOVA — [p-value comment as in outcome 17, analysis 9]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.8 to 0.8]

23. Secondary Outcome: Percent Change From Baseline in Serum Calcium at Weeks 12, 32, 56, and 80
Description: Blood was taken for measurement of serum calcium. Percent change from baseline was based on log transformed data. Geometric mean, GM; standard error, SE. This outcome measure was analyzed for a subset of participants in the bone study only. n is the number of evaluable participants, which is the number of participants with a value at baseline and at the specified visit for the parameter of interest.
Time Frame: Baseline and Weeks 12, 32, 56, and 80
Population: Week 20 Evaluable for the Bone Sub-study Population. This is a subset of the bone sub-study with LOCF from Week 20. Only participants with serum calcium measurements at Week 20 or later were included.
Measure: Number; unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 79 | 79
percent change
  Wk80 % change + SE, overall n= 79, 79 | 0.929 | 1.104
  Wk80 % change, overall n=79, 79 | 0.424 | 0.592
  Wk80 % change - SE, overall n= 79, 79 | -0.079 | 0.083
  Wk56 % change + SE, overall n= 79, 79 | 1.098 | 1.313
  Wk56 % change, overall n= 79, 79 | 0.527 | 0.735
  Wk56 % change - SE, overall n 79, 79 | -0.040 | 0.160
  Wk32 % change + SE, overall n=78, 77 | 0.136 | -0.735
  Wk32 % change, overall n= 78, 77 | -0.316 | -1.204
  Wk32 % change - SE, overall n 78, 79 | -0.766 | -1.607
  Wk12 % change + SE, overall n=81, 78 | 0.568 | -0.315
  Wk12 % change, overall n= 81, 78 | 0.123 | -0.767
  Wk12 % change - SE, overall n 81, 78 | -0.320 | -1.216
  Wk80 % change + SE, males n=34, 39 | 0.8777 | 1.551
  Wk80 % change, males n= 34, 39 | 0.071 | 0.817
  Wk80 % change - SE, males n 34, 39 | -0.728 | 0.877
  Wk56 % change + SE, males n=34, 39 | 1.304 | 1.092
  Wk56 % change, males n= 34, 39 | 0.646 | 0.498
  Wk56 % change - SE, males n 34, 39 | -0.009 | -0.094
  Wk32 % change + SE, males n=33, 39 | -0.538 | -0.585
  Wk32 % change, males n= 33, 39 | -1.281 | -1.254
  Wk32 % change - SE, males n 33,39 | -2.019 | -1.919
  Wk12 % change + SE, males n=37, 40 | 1.410 | 0.543
  Wk12 % change, males n= 37, 40 | 0.656 | -0.147
  Wk12 % change - SE, males n 37, 40 | -0.091 | -0.833
  Wk80 % change + SE, females n= 45, 40 | 1.508 | 1.049
  Wk80 % change, females n=45, 40 | 0.735 | 0.279
  Wk80 % change - SE, females n= 45, 40 | -0.033 | -0.484
  Wk56 % change + SE, females n= 45, 40 | 1.692 | 1.884
  Wk56 % change, females n=45, 40 | 0.720 | 0.911
  Wk56 % change - SE, females n= 45, 40 | -0.242 | -0.053
  Wk32 % change + SE, females n= 45, 38 | 0.637 | -0.653
  Wk32 % change, females n=45, 38 | 0.038 | -1.293
  Wk32 % change - SE, females n= 45, 38 | -0.557 | -1.930
  Wk12 % change + SE, females n= 44, 38 | 0.715 | -0.425
  Wk12 % change, females n=44, 38 | 0.055 | -1.081
  Wk12 % change - SE, females n= 44, 38 | -0.600 | -1.733
  Wk80 % change + SE, premenopausal females n=19, 14 | 1.429 | 0.704
  Wk80 % change, premenopausal females n= 19, 14 | 0.531 | -0.111
  Wk80 % change - SE, premenopausal females n 19, 14 | -0.359 | -0.918
  Wk56 % change + SE, premenopausal females n=19, 14 | 2.091 | 2.334
  Wk56 % change, premenopausal females n= 19, 14 | 0.960 | 1.298
  Wk56 % change - SE, premenopausal females n 19, 14 | -0.159 | 0.273
  Wk32 % change + SE, premenopausal females n=19, 13 | 1.074 | -0.650
  Wk32 % change, premenopausal females n= 19, 13 | 0.070 | -1.679
  Wk32 % change - SE, premenopausal females n 19, 13 | -0.923 | -2.698
  Wk12 % change + SE, premenopausal females n=19, 13 | 0.420 | -0.218
  Wk12 % change, premenopausal females n= 19, 13 | -0.657 | -1.280
  Wk12 % change - SE, premenopausal females n 19, 13 | -1.722 | -2.330
  Wk80 % change+ SE, postmenopausal females n=26, 26 | 2.019 | 1.915
  Wk80 % change, postmenopausal females n=26, 26 | 0.760 | 0.604
  Wk80% change - SE, postmenopausal females n=26, 26 | -0.484 | -0.690
  Wk56 % change+ SE, postmenopausal females n=26, 26 | 2.181 | 2.691
  Wk56 % change, postmenopausal females n=26, 26 | 0.560 | 0.993
  Wk56% change - SE, postmenopausal females n=26, 26 | -1.035 | -0.677
  Wk32 % change+ SE, postmenopausal females n=26, 25 | 0.844 | -0.535
  Wk32 % change, postmenopausal females n=26, 25 | 0.056 | -1.360
  Wk32% change - SE, postmenopausal females n=26, 25 | -0.726 | -2.178
  Wk12 % change+ SE, postmenopausal females n=25, 25 | 0.844 | -1.163
  Wk12 % change, postmenopausal females n=25, 25 | -0.042 | -2.074
  Wk12% change - SE, postmenopausal females n=25, 25 | -0.921 | -2.976
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.7895, ANCOVA — Overall population, Week 80. Log transformed. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 0.168, 95% CI 2-sided [-1.066 to 1.417]
Statistical Analysis 2: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.4155, ANCOVA — Males, Week 80. Log transformed. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 0.745, 95% CI 2-sided [-1.064 to 2.587]
Statistical Analysis 3: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.6223, ANCOVA — Females, Week 80. Log transformed. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = -0.452, 95% CI 2-sided [-2.253 to 1.382]
Statistical Analysis 4: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.5908, ANCOVA — Premenopausal females, Week 80. Log transformed. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = -0.638, 95% CI 2-sided [-3.043 to 1.826]
Statistical Analysis 5: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.9154, ANCOVA — Postmenopausal females, Week 80. Log transformed. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = -0.155, 95% CI 2-sided [-3.037 to 2.814]

24. Secondary Outcome: Percent Change From Baseline in Intact Parathyroid Hormone at Week 80
Description: Blood was taken for measurement of intact parathyroid hormone. Percent change from baseline was based on log transformed data. Standard error, SE; Wk, Week; %, percent. This outcome measure was analyzed for a subset of participants in the bone study only. n is the number of evaluable participants, which is the number of participants with a value at baseline and at the specified visit for the parameter of interest.
Time Frame: Baseline and Week 80
Population: Week 20 Evaluable for the Bone Sub-study Population. This is a subset of the bone sub-study with LOCF from Week 20. Only participants with intact parathyroid hormone measurements at Week 20 or later were included.
Measure: Number; unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 45 | 38
percent change
  Wk80 % change + SE, overall n= 45, 38 | -1.296 | 0.843
  Wk80 % change, overall n=45, 38 | -7.634 | -6.279
  Wk80 % change - SE, overall n= 45, 38 | -13.565 | -12.898
  Wk80 % change + SE, males n=16, 21 | -1.160 | -2.619
  Wk80 % change, males n= 16, 21 | -9.238 | -8.941
  Wk80 % change - SE, males n=16, 21 | -16.655 | -14.852
  Wk80 % change + SE, females n= 30, 22 | 4.662 | 11.166
  Wk80 % change, females n=30, 22 | -4.608 | -1.759
  Wk 80 % change - SE, females n= 30, 22 | -13.056 | -13.182
  Wk80 % change + SE, premenopausal females n=13, 7 | 14.295 | 24.396
  Wk80 % change, premenopausal females n= 13, 7 | -7.686 | -0.126
  Wk80 % change - SE, premenopausal females n=13, 7 | -25.440 | -20.160
  Wk80 % change+ SE, postmenopausal females n=16, 10 | 3.017 | 8.297
  Wk80 % change, postmenopausal females n=16, 10 | -12.109 | -9.170
  Wk80% change - SE, postmenopausal females n=16, 10 | -25.014 | -23.807
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.8682, ANCOVA — Overall population, Week 80. Log transformed; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 1.467, 95% CI 2-sided [-14.785 to 20.818]
Statistical Analysis 2: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.9740, ANCOVA — Males, Week 80. Log transformed; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 0.328, 95% CI 2-sided [-18.308 to 23.214]
Statistical Analysis 3: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.8378, ANCOVA — Females, Week 80. Log transformed; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 2.986, 95% CI 2-sided [-22.997 to 37.735]
Statistical Analysis 4: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.7889, ANCOVA — Pre-menopausal females, Week 80. Log transformed; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 8.190, 95% CI 2-sided [-43.839 to 108.422]
Statistical Analysis 5: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.8800, ANCOVA — Postmenopausal females, Week 80. Log transformed; .Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 3.344, 95% CI 2-sided [-34.853 to 63.935]

25. Secondary Outcome: Percent Change From Baseline in 25-hydroxy Vitamin D at Week 80
Description: Blood was taken for measurement of 25-hydroxy vitamin D. Percent change from baseline was based on log transformed data. Standard error, SE; Wk, Week; %, percent. This outcome measure was analyzed for a subset of participants in the bone study only. n is the number of evaluable participants, which is the number of participants with a value at baseline and at the specified visit for the parameter of interest.
Time Frame: Baseline and Week 80
Population: Week 20 Evaluable for the Bone Sub-study Population. This is a subset of the bone sub-study with LOCF from Week 20. Only participants with 25-hydroxy vitamin D measurements at Week 20 or later were included.
Measure: Number; unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 45 | 38
percent change
  Wk80 % change + SE, overall n= 45, 38 | -7.0053 | -4.6305
  Wk80 % change, overall n=45, 38 | -13.9678 | -12.9210
  Wk 80 % change - SE, overall n= 45, 38 | -20.4091 | -20.4909
  Wk80 % change + SE, males n=16, 21 | 8.9639 | -4.2837
  Wk80 % change, males n=16, 21 | -4.4369 | -14.1507
  Wk80 % change - SE, males n=16, 21 | -16.1896 | -23.0005
  Wk80 % change + SE, females n= 29, 17 | -7.1080 | 4.7124
  Wk80 % change, females n=29, 17 | -16.4578 | -9.0412
  Wk 80 % change - SE, females n= 29, 17 | -24.8664 | -20.9882
  Wk80 % change + SE, premenopausal females n=13, 7 | -2.0833 | 0.3546
  Wk80 % change, premenopausal females n= 13, 7 | -15.3838 | -16.2325
  Wk80 % change - SE, premenopausal females n=13, 7 | -26.8776 | -30.0781
  Wk80 % change+ SE, postmenopausal females n=16, 10 | 8.8368 | 17.3807
  Wk80 % change, postmenopausal females n=16, 10 | -7.1318 | -2.7100
  Wk80% change - SE, postmenopausal females n=16, 10 | -20.7575 | -19.3620
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.9069, ANCOVA — Overall population, Week 80. Log transformed; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 1.2168, 95% CI 2-sided [-17.6057 to 24.3392]
Statistical Analysis 2: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.5118, ANCOVA — Males, Week 80. Log transformed; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = -10.1648, 95% CI 2-sided [-35.6298 to 25.3742]
Statistical Analysis 3: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.5816, ANCOVA — Females, Week 80. Log transformed; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 8.8777, 95% CI 2-sided [-20.2636 to 48.6692]
Statistical Analysis 4: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.9587, ANCOVA — Pre-menopausal females, Week 80. Log transformed; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = -1.0031, 95% CI 2-sided [-35.9280 to 52.9590]
Statistical Analysis 5: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.8337, ANCOVA — Postmenopausal females, Week 80. Log transformed; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 4.7614, 95% CI 2-sided [-34.4741 to 67.4901]

26. Secondary Outcome: Percent Change From Baseline in Estradiol at Weeks 20, 56, and 80
Description: Blood was taken for measurement of estradiol. Percent change from baseline was based on log transformed data. Standard error, SE; Wk, Week; %, percent. This outcome measure was analyzed for a subset of female participants in the bone study only. n is the number of evaluable participants, which is the number of female participants with a value at baseline and at the specified visit for the parameter of interest.
Time Frame: Baseline and Weeks 20, 56, and 80
Population: Week 20 Evaluable for the Bone Sub-study Population. This is a subset of the bone sub-study with LOCF from Week 20. Only participants with estradiol measurements at Week 20 or later were included.
Measure: Number; unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 30 | 22
percent change
  Wk80 % change + SE, females n= 30, 22 | -8.695 | 0.097
  Wk80 % change, females n=30, 22 | -21.360 | -15.441
  Wk 80 % change - SE, females n= 30, 22 | -32.268 | -28.567
  Wk56 % change + SE, females n= 27, 21 | 12.015 | 10.268
  Wk56 % change, females n=27, 21 | -0.815 | -2.439
  Wk 56 % change - SE, females n= 27, 21 | -12.175 | -13.682
  Wk20 % change + SE, females n= 36, 25 | 7.863 | 14.875
  Wk20 % change, females n=36, 25 | -5.097 | -0.646
  Wk 20 % change - SE, females n= 36, 25 | -16.500 | -14.875
  Wk80 % change + SE, premenopausal females n=13, 9 | 25.386 | 67.328
  Wk80 % change, premenopausal females n= 13, 9 | -17.314 | 7.667
  Wk80 % change - SE, premenopausal females n=13, 9 | -45.472 | -30.722
  Wk56 % change + SE, premenopausal females n=12, 8 | 35.708 | 19.557
  Wk56 % change, premenopausal females n= 12, 8 | 1.677 | -11.431
  Wk56 % change - SE, premenopausal females n=12, 8 | -23.820 | -34.386
  Wk20 % change + SE, premenopausal females n=15, 10 | 5.738 | 8.866
  Wk20 % change, premenopausal females n=15, 10 | -3.721 | -3.005
  Wk20 % change - SE, premenopausal females n=15, 10 | -12.334 | -13.581
  Wk80 % change+ SE, postmenopausal females n=17, 13 | -27.303 | -25.501
  Wk80 % change, postmenopausal females n=17, 13 | -33.045 | -31.754
  Wk80% change - SE, postmenopausal females n=17, 13 | -38.334 | -37.482
  Wk56 % change+ SE, postmenopausal females n=15, 13 | -25.758 | -18.475
  Wk56 % change, postmenopausal females n=15, 13 | -32.766 | -25.372
  Wk56% change - SE, postmenopausal females n=15, 13 | -39.113 | -31.686
  Wk20 % change+ SE, postmenopausal females n=21, 15 | 3.432 | 16.140
  Wk20 % change, postmenopausal females n=21, 15 | -12.870 | -5.061
  Wk20% change - SE, postmenopausal females n=21, 15 | -26.603 | -22.391
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.7041, ANCOVA — [p-value comment as in outcome 23, analysis 3]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 7.527, 95% CI 2-sided [-26.773 to 57.892]
Statistical Analysis 2: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.6403, ANCOVA — Pre-menopausal females, Week 80. Log transformed. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 30.211, 95% CI 2-sided [-61.586 to 341.371]
Statistical Analysis 3: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.8474, ANCOVA — [p-value comment as in outcome 23, analysis 5]; .Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 1.929, 95% CI 2-sided [-17.015 to 25.198]

27. Secondary Outcome: Percent Change From Baseline in C-terminal Telopeptide (CTX) at Weeks 20, 56, and 80
Description: Blood was taken for measurement of CTX. Percent change from baseline was based on log transformed data. Standard error, SE; Wk, Week; %, percent. This outcome measure was analyzed for a subset of participants in the bone study only. n is the number of evaluable participants, which is the number of participants with a value at baseline and at the specified visit for the parameter of interest.
Time Frame: Baseline and Weeks 20, 56, and 80
Population: Week 20 Evaluable for the Bone Sub-study Population. This is a subset of the bone sub-study with LOCF from Week 20. Only participants with CTX measurements at Week 20 or later were included.
Measure: Number; unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 69 | 62
percent change
  Wk80 % change + SE, overall n=69, 62 | -12.7 | -7.5
  Wk80 % change, overall n=69, 62 | -18.7 | -14.0
  Wk80 % change - SE, overall n=79, 62 | -24.2 | -20.1
  Wk56 % change + SE, overall n=68, 62 | -5.3 | 3.7
  Wk56 % change, overall n=68, 62 | -11.4 | -3.2
  Wk56 % change - SE, overall n=68, 62 | -17.1 | -9.6
  Wk20 % change + SE, overall n=61, 56 | -0.8 | -0.8
  Wk20 % change, overall n=61, 56 | -5.5 | -5.9
  Wk20 % change - SE, overall n=61, 56 | -9.9 | -10.7
  Wk80 % change + SE, males n=28, 32 | -11.0 | -1.8
  Wk80 % change, males n=28, 32 | -20.7 | -10.9
  Wk80 % change - SE, males n=28, 32 | -29.2 | -19.1
  Wk56 % change + SE, males n=28, 32 | -11.5 | 6.5
  Wk56 % change, males n=28, 32 | -20.0 | -2.2
  Wk56 % change - SE, males n=28, 32 | -27.7 | -10.2
  Wk20 % change + SE, males n=23, 29 | 4.8 | 13.2
  Wk20 % change, males n=23, 29 | -3.1 | 5.8
  Wk20 % change - SE, males n=23, 29 | -10.3 | -1.1
  Wk80 % change + SE, females n=41, 30 | -12.9 | -8.2
  Wk80 % change, females n=41, 30 | -20.1 | -16.9
  Wk80 % change - SE, females n=41, 30 | -26.6 | -24.8
  Wk56 % change + SE, females n=40, 30 | -8.5 | 1.2
  Wk56 % change, females n=40, 30 | -15.8 | -8.0
  Wk56 % change - SE, females n=40, 30 | -22.5 | -16.4
  Wk20 % change + SE, females n=38, 27 | -2.5 | -8.3
  Wk20 % change, females n=38, 27 | -8.9 | -15.3
  Wk20 % change - SE, females n=38, 27 | -15.0 | -21.7
  Wk80 % change + SE, premenopausal females n=18, 9 | -18.6 | 10.9
  Wk80 % change, premenopausal females n=18, 9 | -27.8 | -4.7
  Wk80 % change - SE, premenopausal females n=18, 9 | -36.0 | -18.1
  Wk56 % change + SE, premenopausal females n=18, 9 | -25.5 | 12.6
  Wk56 % change, premenopausal females n=18, 9 | -31.8 | 0.8
  Wk56 % change - SE, premenopausal females n=18, 9 | -37.5 | -9.8
  Wk20 % change + SE, premenopausal females n=16, 9 | -4.2 | -7.8
  Wk20 % change, premenopausal females n=16, 9 | -14.0 | -18.9
  Wk20 % change - SE, premenopausal females n=16, 9 | -22.8 | -28.8
  Wk80 % change+ SE, postmenopausal females n=23, 21 | -11.5 | -14.3
  Wk80 % change, postmenopausal females n=23, 21 | -21.0 | -24.4
  Wk80% change - SE, postmenopausal females n=23, 21 | -29.5 | -33.4
  Wk56 % change+ SE, postmenopausal females n=22, 21 | 10.3 | 5.1
  Wk56 % change, postmenopausal females n=22, 21 | -2.1 | -7.4
  Wk56% change - SE, postmenopausal females n=22, 21 | -13.0 | -18.4
  Wk20 % change+ SE, postmenopausal females n=22, 18 | 4.1 | -3.2
  Wk20 % change, postmenopausal females n=22, 18 | -5.8 | -13.6
  Wk20% change - SE, postmenopausal females n=22, 18 | -14.7 | -22.8
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.4860, ANCOVA — Overall, Week 80. Log transformed. If the p value was significant at Week 80 a comparison was done at Week 56; if it was significant at Weeks 80 and 56, a comparison was done at Week 20; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 5.7, 95% CI 2-sided [-9.6 to 23.6]
Statistical Analysis 2: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.3791, ANCOVA — [p-value comment as in outcome 23, analysis 2]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 12.3, 95% CI 2-sided [-13.7 to 46.1]
Statistical Analysis 3: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.7065, ANCOVA — [p-value comment as in outcome 23, analysis 3]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 4.0, 95% CI 2-sided [-15.3 to 27.6]
Statistical Analysis 4: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.1381, ANCOVA — [p-value comment as in outcome 26, analysis 2]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 32.1, 95% CI 2-sided [-9.5 to 92.7]
Statistical Analysis 5: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.7195, ANCOVA — [p-value comment as in outcome 23, analysis 5]; .Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = -4.3, 95% CI 2-sided [-25.4 to 22.7]

28. Secondary Outcome: Percent Change From Baseline in Procollagen Type-1 N-propeptide (P1NP) at Weeks 20, 56, and 80
Description: Blood was taken for measurement of P1NP. Percent change from baseline was based on log transformed data. Standard error, SE; Wk, Week; %, percent. This outcome measure was analyzed for a subset of participants in the bone study only. n is the number of evaluable participants, which is the number of participants with a value at baseline and at the specified visit for the parameter of interest.
Time Frame: Baseline and Weeks 20, 56, and 80
Population: Week 20 Evaluable for the Bone Sub-study Population. This is a subset of the bone sub-study with LOCF from Week 20. Only participants with P1NP measurements at Week 20 or later were included.
Measure: Number; unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 72 | 64
percent change
  Wk80 % change + SE, overall n= 72, 64 | -18.4 | -20.7
  Wk80 % change, overall n=72, 64 | -22.0 | -24.3
  Wk80 % change - SE, overall n=72, 64 | -25.5 | -27.8
  Wk56 % change + SE, overall n=72, 64 | -23.5 | -26.6
  Wk56 % change, overall n=72, 64 | -26.9 | -30.0
  Wk56 % change - SE, overall n=72, 64 | -30.2 | -33.3
  Wk20 % change + SE, overall n=66, 59 | -24.0 | -31.6
  Wk20 % change, overall n=66, 59 | -27.0 | -34.6
  Wk20 % change - SE, overall n=66, 59 | -30.0 | -37.5
  Wk80 % change + SE, males n=30, 32 | -18.5 | -18.2
  Wk80 % change, males n=30, 32 | -24.1 | -23.4
  Wk80 % change - SE, males n=30, 32 | -29.4 | -28.2
  Wk56 % change + SE, males n=30, 32 | -22.7 | -23.0
  Wk56 % change, males n=30, 32 | -27.7 | -27.6
  Wk56 % change - SE, males n=30, 32 | -32.4 | -31.9
  Wk20 % change + SE, males n=26, 29 | -20.2 | -24.7
  Wk20 % change, males n=26, 29 | -25.4 | -29.5
  Wk20 % change - SE, males n=26, 29 | -30.3 | -33.9
  Wk80 % change + SE, females n=42, 32 | -19.3 | -19.2
  Wk80 % change, females n=42, 32 | -23.8 | -24.4
  Wk80 % change - SE, females n=42, 32 | -28.2 | -29.3
  Wk56 % change + SE, females n=42, 32 | -28.6 | -27.0
  Wk56 % change, females n=42, 32 | -32.8 | -32.0
  Wk56 % change - SE, females n=42, 32 | -36.9 | -36.6
  Wk20 % change + SE, females n=40, 30 | -25.2 | -31.6
  Wk20 % change, females n=40, 30 | -30.0 | -36.6
  Wk20 % change - SE, females n=40, 30 | -34.5 | -41.2
  Wk80 % change + SE, premenopausal females n=19, 10 | -16.9 | -11.0
  Wk80 % change, premenopausal females n=19, 10 | -23.6 | -20.1
  Wk80 % change - SE, premenopausal females n=19, 10 | -29.7 | -28.3
  Wk56 % change + SE, premenopausal females n=19, 10 | -25.3 | -23.4
  Wk56 % change, premenopausal females n=19, 10 | -31.0 | -30.9
  Wk56 % change - SE, premenopausal females n=19, 10 | -36.2 | -37.6
  Wk20 % change + SE, premenopausal females n=17, 10 | -24.6 | -29.0
  Wk20 % change, premenopausal females n=17, 10 | -31.4 | -36.5
  Wk20 % change - SE, premenopausal females n=17, 10 | -37.7 | -43.1
  Wk80 % change+ SE, postmenopausal females n=23, 22 | -22.5 | -27.6
  Wk80 % change, postmenopausal females n=23, 22 | -28.4 | -33.8
  Wk80% change - SE, postmenopausal females n=23, 22 | -33.8 | -39.4
  Wk56 % change+ SE, postmenopausal females n=23, 22 | -32.1 | -35.2
  Wk56 % change, postmenopausal females n=23, 22 | -37.9 | -41.4
  Wk56% change - SE, postmenopausal females n=22, 22 | -43.2 | -47.0
  Wk20 % change+ SE, postmenopausal females n=23, 20 | -25.2 | -34.0
  Wk20 % change, postmenopausal females n=23, 20 | -31.9 | -40.9
  Wk20% change - SE, postmenopausal females n=23, 20 | -38.0 | -47.1
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.5595, ANCOVA — [p-value comment as in outcome 27, analysis 1]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = -3.0, 95% CI 2-sided [-12.3 to 7.4]
Statistical Analysis 2: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.9125, ANCOVA — [p-value comment as in outcome 23, analysis 2]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 1.0, 95% CI 2-sided [-15.3 to 20.4]
Statistical Analysis 3: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.9122, ANCOVA — [p-value comment as in outcome 23, analysis 3]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = -0.8, 95% CI 2-sided [-14.0 to 14.5]
Statistical Analysis 4: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.7435, ANCOVA — [p-value comment as in outcome 26, analysis 2]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 4.6, 95% CI 2-sided [-21.2 to 38.7]
Statistical Analysis 5: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.3897, ANCOVA — [p-value comment as in outcome 23, analysis 5]; .Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = -7.5, 95% CI 2-sided [-23.0 to 11.0]

29. Secondary Outcome: Percent Change From Baseline in Bone Alkaline Phosphatase (BSAP) at Weeks 20, 56, and 80
Description: Blood was taken for measurement of BSAP. Percent change from baseline was based on log transformed data. Standard error, SE; Wk, Week; %, percent. This outcome measure was analyzed for a subset of participants in the bone study only. n is the number of evaluable participants, which is the number of participants with a value at baseline and at the specified visit for the parameter of interest.
Time Frame: Baseline and Weeks 20, 56, and 80
Population: Week 20 Evaluable for the Bone Sub-study Population. This is a subset of the bone sub-study with LOCF from Week 20. Only participants with BSAP measurements at Week 20 or later were included.
Measure: Number; unit: percent change
Arm/Group | Metformin | Avandamet
Number analyzed (Participants) | 72 | 64
percent change
  Wk80 % change + SE, overall n=72, 64 | -21.19 | -23.30
  Wk80 % change, overall n=72, 64 | -24.23 | -26.37
  Wk80 % change - SE, overall n=72, 64 | -27.15 | -29.31
  Wk56 % change + SE, overall n=72, 64 | -18.29 | -24.39
  Wk56 % change, overall n=72, 64 | -21.52 | -27.48
  Wk56 % change - SE, overall n=72, 64 | -24.61 | -30.45
  Wk20 % change + SE, overall n=66, 59 | -24.16 | -31.02
  Wk20 % change, overall n=66, 59 | -26.46 | -33.31
  Wk20 % change - SE, overall n=66, 59 | -28.70 | -35.53
  Wk80 % change + SE, males n=30, 32 | -15.44 | -21.18
  Wk80 % change, males n=30, 32 | -20.35 | -25.34
  Wk80 % change - SE, males n=30, 32 | -24.97 | -29.27
  Wk56 % change + SE, males n=30, 32 | -12.22 | -21.97
  Wk56 % change, males n=30, 32 | -17.05 | -25.87
  Wk56 % change - SE, males n=30, 32 | -21.62 | -29.57
  Wk20 % change + SE, males n=26, 29 | -16.27 | -26.59
  Wk20 % change, males n=26, 29 | -20.50 | -30.05
  Wk20 % change - SE, males n=26, 29 | -24.51 | -33.35
  Wk80 % change + SE, females n=42, 32 | -24.30 | -23.20
  Wk80 % change, females n=42, 32 | -28.11 | -27.60
  Wk80 % change - SE, females n=42, 32 | -31.74 | -31.74
  Wk56 % change + SE, females n=42, 32 | -22.54 | -24.09
  Wk56 % change, females n=42, 32 | -26.75 | -28.77
  Wk56 % change - SE, females n=42, 32 | -30.73 | -33.17
  Wk20 % change + SE, females n=40, 30 | -26.82 | -31.60
  Wk20 % change, females n=40, 30 | -30.23 | -35.23
  Wk20 % change - SE, females n=40, 30 | -33.48 | -38.66
  Wk80 % change + SE, premenopausal females n=19, 10 | -13.89 | -23.69
  Wk80 % change, premenopausal females n=19, 10 | -19.28 | -29.89
  Wk80 % change - SE, premenopausal females n=19, 10 | -24.33 | -35.59
  Wk56 % change + SE, premenopausal females n=19, 10 | -12.43 | -27.74
  Wk56 % change, premenopausal females n=19, 10 | -16.84 | -32.47
  Wk56 % change - SE, premenopausal females n=19, 10 | -21.02 | -36.89
  Wk20 % change + SE, premenopausal females n=17, 10 | -24.73 | -32.69
  Wk20 % change, premenopausal females n=17, 10 | -29.57 | -37.68
  Wk20 % change - SE, premenopausal females n=17, 10 | -34.10 | -42.32
  Wk80 % change+ SE, postmenopausal females n=23, 22 | -29.10 | -25.82
  Wk80 % change, postmenopausal females n=23, 22 | -34.39 | -31.93
  Wk80% change - SE, postmenopausal females n=23, 22 | -39.29 | -37.54
  Wk56 % change+ SE, postmenopausal females n=23, 22 | -27.51 | -23.61
  Wk56 % change, postmenopausal females n=23, 22 | -34.04 | -31.20
  Wk56% change - SE, postmenopausal females n=23, 22 | -39.99 | -38.04
  Wk20 % change+ SE, postmenopausal females n=23, 20 | -28.14 | -32.02
  Wk20 % change, postmenopausal females n=23, 20 | -32.70 | -36.94
  Wk20% change - SE, postmenopausal females n=23, 20 | -36.97 | -41.50
Statistical Analysis 1: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.5176, ANCOVA — [p-value comment as in outcome 27, analysis 1]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = -2.83, 95% CI 2-sided [-10.97 to 6.06]
Statistical Analysis 2: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.3620, ANCOVA — [p-value comment as in outcome 23, analysis 2]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = -6.26, 95% CI 2-sided [-18.62 to 7.97]
Statistical Analysis 3: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.9115, ANCOVA — [p-value comment as in outcome 23, analysis 3]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 0.72, 95% CI 2-sided [-11.39 to 14.48]
Statistical Analysis 4: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.1956, ANCOVA — [p-value comment as in outcome 26, analysis 2]; Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = -13.51, 95% CI 2-sided [-30.35 to 8.31]
Statistical Analysis 5: Comparison: Metformin vs Avandamet; Test type: Superiority or Other; p = 0.6749, ANCOVA — [p-value comment as in outcome 23, analysis 5]; .Based on ANCOVA with terms for treatment, region, pre-screening HbA1c strata, sex, baseline; Percent difference from metformin = 3.75, 95% CI 2-sided [-13.09 to 23.85]

ADVERSE EVENTS:
Time Frame: An on therapy adverse event (AE)/serious adverse event (SAE) was defined as an AE/SAE with onset on or after the start date of study medication but not later than two days after the last date of study medication.
Description: SAEs and AEs were collected in the Safety Population, comprised of all participants who were randomized and received at least one dose of the study medication.
Arm/Group | Metformin | Avandamet
Serious Adverse Events (participants affected / at risk) | 27/334 | 28/344
Other Adverse Events (participants affected / at risk) | 159/334 | 145/344
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=334) | Avandamet (N=344)
Pneumonia (Infections and infestations) | 2 | 2
Appendicitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 2 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Localized infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 9
Coronary artery disease (Cardiac disorders) | 1 | 2
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac discomfort (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Cranial neuropathy (Nervous system disorders) | 1 | 0
Haemorrhage itracranial (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Intrevertebral disc protusion (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1
Angle closure glaucoma (Eye disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=334) | Avandamet (N=344)
Diarrhoea (Gastrointestinal disorders) | 63 | 41
Nausea (Gastrointestinal disorders) | 30 | 31
Upper respiratort tract infection (Infections and infestations) | 30 | 22
Headache (Nervous system disorders) | 26 | 19
Nasopharyngitis (Infections and infestations) | 26 | 18
Dizziness (Nervous system disorders) | 24 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 16
Urinary tract infection (Infections and infestations) | 20 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 25
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 22
Oedema peripheral (General disorders) | 4 | 16

LIMITATIONS AND CAVEATS:
Ten participants who started the study and were randomized did not receive any study medication (6 participants in the metformin arm and 4 participants in the avandamet arm). These participants are not included in any of the analysis populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.